CLINICAL TRIAL: NCT03004131
Title: Clinical Trial to Assess Onset of Action of Azelastine Hydrochloride and Fluticasone Propionate Nasal Spray Delivered in a Single Spray (MP-AzeFlu) in the Treatment of Allergen-Induced Allergic Rhinitis Symptoms in Comparison to Placebo and Free Combination of Fluticasone Propionate Nasal Spray and Oral Loratadine
Brief Title: MP-AzeFlu Allergen Chamber - Onset of Action Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: X-03065-3311
Record Dates: First submitted 2016-12-16; First posted 2016-12-28 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2017-05

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — azelastine; Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fixed drug combination (Experimental): MP29-02 or MP-AzuFlu as fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray (Dymista) plus Placebo tablet
  Interventions: Drug: Azelastine hydrochloride + fluticasone propionate nasal spray
- Placebo (Placebo Comparator): Nasal spray with no active dose plus Placebo tablet
  Interventions: Drug: Placebos
- active control (Active Comparator): fluticasone propionate nasal spray (Flonase) plus loratadine 10 mg tablets (Claritin)
  Interventions: Drug: fluticasone propionate nasal spray + loratadine

INTERVENTIONS:
Drug: Azelastine hydrochloride + fluticasone propionate nasal spray
  Arms: fixed drug combination
Drug: Placebos
  Arms: Placebo
Drug: fluticasone propionate nasal spray + loratadine
  Arms: active control

SUMMARY:
This study is to assess the onset of action of fixed drug combination of azelastine hydrochloride and fluticasone propionate nasal spray (MP-AzeFlu) in treating the nasal symptoms of seasonal allergic rhinitis (SAR) induced by an allergen challenge in an Environmental Exposure Chamber (EEC).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Male or female subjects (childbearing and non-childbearing potential, defined as females with no menstruation for a minimum of 12 months prior to screening) aged 18 to 55 years (inclusive) at screening.
3. History of SAR to ragweed pollen for at least the previous 2 ragweed pollen seasons.
4. Positive skin prick test (SPT) response to ragweed pollen (allergen induced wheal diameter at least 3 mm larger than the negative control). A test performed in the previous 12 months may be used to qualify the subject.

   To be eligible for Visit 2 EEC, a subject must additionally comply with the following criteria:
5. Asymptomatic or with mild symptoms during the baseline recording of symptoms prior to start of the screening EEC (Visit 2):

   - TNSS ≤ 3/12 with the score for each symptom being less than 2.

   To be eligible for Visit 3, a subject must additionally comply with the following criteria during Visit 2 EEC:
6. Demonstrate adequate symptomology:

   - TNSS ≥ 6/12 on at least two ePDAT™ time point assessments during hours 0-2 in the EEC (Visit 2), with at least one occurring during the last two time points. Additionally, subjects will be required to meet a score of at least 2/3 for runny nose at least twice during hours 0-2 in the EEC, with at least one occurring during the last two time points.

   To be eligible for randomisation (Visit 3), a subject must additionally comply with the following criteria:
7. Demonstrate adequate symptomology:

   * TNSS ≥ 6/12 on at least two ePDAT™ time point assessments during hours 0-2 in the EEC (Visit 3), with at least one occurring during the last two time points. Additionally, subjects will be required to meet a score of at least 2/3 for runny nose at least twice during hours 0-2 in the EEC, with at least one occurring during the last two time points.
   * No evidence of complete nasal blockage on either one or both sides on anterior rhinoscopy within 30 minutes prior to dosing.

Exclusion Criteria:

Safety concerns:

1. History of allergic reaction to fluticasone propionate, azelastine hydrochloride, loratadine, or one of the excipients of the study treatments (e.g. benzalkonium chloride, phenylethyl alcohol, microcrystalline cellulose) or a component of the container.
2. History of anaphylaxis, cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, metabolic, psychiatric, neurological, or other disease at screening that may affect subject safety during the study or evaluation of the study endpoints at the discretion of the Investigator and/or designee.
3. Subjects with a current diagnosis of asthma or subjects with measured FEV1 <75% of the predicted value.
4. Pregnant, breast-feeding or planning a pregnancy during the study and women of childbearing potential not using adequate contraception. Women of childbearing potential not abstinent or using a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs, tubal ligation or vasectomised partner started at least 4 weeks prior to screening.

   Lack of suitability for the study:
5. Previous and concomitant treatments: use of prohibited therapies (Antihistaminic agents,Theophylline, Cromolyn sodium, Corticosteroids, Decongestants, Immunotherapy, Systemic antibiotics, any cytochrome P450 3A4 inhibiting or inducing drug [e.g. ritonavir, ketoconazole, itraconazole, erythromycin, cimetidine, rifampicin, St. John's wort (Hypericum perforatum) etc.], Tricyclic antidepressants and MAO inhibitors ); and use of any medication considered to have an influence on the outcome of the study during the EEC session, at the discretion of the Investigator and/or designee.
6. Subjects with (expected) clinically relevant symptoms at the timing of the scheduled EEC assessments due to concomitant sensitization, i.e., positive SPT (mean wheal diameter at least 3 mm larger than the negative control) and a history of allergic response to the causative allergen, at the discretion of the Investigator. Subjects with a positive SPT for cats and/or dogs are acceptable if the subject avoids cats and/or dogs for the duration of the study.
7. Concomitant diseases: abnormalities during the screening visit that might interfere with study results as determined by the Investigator and/or designee.
8. Presence of a severely deviated septum, septal perforation, structural nasal defect or large nasal polyps causing obstruction as determined by the Investigator.
9. Acute conditions: any acute illness within 7 days prior to the screening visit, including acute conjunctivitis or any other ocular infection.
10. History of increased ocular pressure, glaucoma and/or cataracts.
11. Tuberculosis, untreated local or systemic fungal or bacterial infections, systemic viral or parasitic infections or ocular herpes simplex.
12. Recent nasal ulcers, mucosal erosion, nasal surgery, or nasal trauma, as judged by the Investigator.
13. Exposure to chickenpox or measles within 4 weeks prior to the screening visit or during the study.
14. History of chronic sinusitis or history of non-allergic rhinitis.
15. Exposure to another investigational product within the last 30 days prior to screening.
16. History of malignancy within the past five years, except for basal cell skin carcinomas that have been treated with no recurrence for at least 3 months.
17. Neurological or psychiatric disease or drug or alcohol abuse which would interfere with the subject's proper completion of the protocol assignment. Subjects with a positive urine drug screen will be excluded.
18. Subjects undergoing surgical procedures with general anaesthesia within 90 days prior to screening or who plan to undergo surgery/hospitalization during the study.

    Administrative reasons:
19. Vulnerable subjects (such as persons kept in detention).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2017-01-07 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS); change from baseline over the last 4 hours of exposure in an Environmental Exposure Chamber (EEC) | Onset of action (first significant difference to placebo) up to 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kolb, Study Director — MEDA Pharma GmbH & Co. KG
Locations (1):
- Inflamax Research, Mississauga, Ontario, Canada